CLINICAL TRIAL: NCT06841575
Title: Advancing Pediatric Retinal Imaging With Auto-aligned OCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00116369; R21EY036545 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Eye Diseases; Retinal Disease; Glaucoma; Optic Nerve Diseases
Keywords: Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Eye Diseases; Retinal Diseases; Glaucoma; Optic Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: Healthy adult volunteers (Experimental): Healthy adult volunteers recruited from the patient population, students or employees of Duke University or Duke Eye Center (n=20)
  Interventions: Device: Auto-aligned OCT
- Group 2: Adult patients in ophthalmology clinics (Experimental): Adult participants recruited from the patient population of Duke Eye Center undergoing clinical examination (n=20)
  Interventions: Device: Auto-aligned OCT
- Group 3: Pediatric patients in ophthalmology clinics (Experimental): Minor participants recruited from the patient population of Duke Eye Center undergoing clinical examination (n=10)
  Interventions: Device: Auto-aligned OCT

INTERVENTIONS:
Device: Auto-aligned OCT — Swept Source OCT system with improved hand-held probe technology for auto-alignment to the patient's eye, as well as on-line detection of image quality and auto-saving at the proper time

SUMMARY:
The goal of the current study is to conduct a pilot study to test a new version of the handheld OCT device capable of auto-alignment to image the retina in adult volunteers, and adult and pediatric patients in clinic.

DETAILED DESCRIPTION:
Handheld OCT imaging is an advancement in ophthalmic imaging technology allowing us to image the pediatric retina. lt has tremendous potential to be applied to assess the structure and blood flow of children with retinal vascular diseases or as a screening tool for pediatric retinal diseases. Despite progress in the development of hand-held OCT probes, there remains a critical gap in technology to achieve fast, proper alignment between the imaging device and the infant eye. Even with the most skilled operators, to acquire consistent OCT and OCTA data capture for longitudinal follow up in uncooperative patients at the bedside remains difficult. lmprovements in hand-held OCT probe technology for auto-alignment to the patient's eye, as well as on-line detection of image quality and auto-saving at the proper time, would address this critical gap in handheld OCT technology. Our biomedical engineering team, has developed prior iterations of the handheld OCT devices and successfully imaged the pediatric retina. The goal of the current study is to conduct a pilot study to test a new version of the handheld OCT device capable of auto-alignment to image the retina in adult volunteers, and adult and pediatric patients in clinic.

The investigators plan to enroll 20 healthy adult volunteers, 20 adult patients and 10 pediatric patients from the ophthalmology clinic. This is an observational study. There are no known risks associated with handheld OCT imaging and no adverse events identified imaging with prior iterations of handheld OCT devices. lmaging data will be downloaded to a secure server for protocol image processing, segmentation, and analysis per protocol in the Duke Advanced Research in SS/SDOCT lmaging (DARSI) laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Healthy adult volunteers
* Subject is able and willing to consent to study participation
* Subject is more than 18 years of age
* Healthy adult volunteers without known ocular issues other than refractive error
* Group 2: Adult patients in ophthalmology clinics
* Health care provider, knowledgeable of protocol, agrees that study personnel could contact the subject
* Subject is able and willing to consent to study participation
* Subject is more than 18 years of age and is a patient in the Duke Eye Center ophthalmology clinics
* Group 3: Pediatric participants in ophthalmology clinics
* Health care provider, knowledgeable of protocol, agrees that study personnel could contact the parent/legal guardian
* Parent/legal guardian is able and willing to consent to study participation
* Pediatric patient less than 18 years of age in Duke Eye Center ophthalmology clinics or undergoing clinically-indicated examination under anesthesia at Duke Eye Center

Exclusion Criteria:

* Group 1: Healthy adult volunteers
* Students or employees under direct supervision of the investigators
* Subjects with prior problems with pupil dilation
* Pregnant woman if receiving dilating drops
* Group 2: Adult patients in ophthalmology clinics
* Participant has a health or eye condition that preclude eye examination or retinal imaging (such as corneal opacity or cataract)
* Group 3: Pediatric participants in ophthalmology clinics
* Parent/legal guardian unwilling or unable to provide consent
* Participant has a health or eye condition that preclude eye examination or retinal imaging (such as corneal opacity or cataract)

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with abnormal retinal microanatomy | Up to 4 single imaging sessions at clinical visits over 2 years
  Measured by optical coherence tomography (OCT) reading.
Severity of abnormal retinal microanatomy | Up to 4 single imaging sessions at clinical visits over 2 years
  Measured by optical coherence tomography (OCT) reading.
Retinal thickness (microns) at the fovea and surrounding optic nerve as measured by OCT analysis | Up to 4 single imaging sessions at clinical visits over 2 years
  Measured by optical coherence tomography (OCT) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Chen, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No